CLINICAL TRIAL: NCT01418105
Title: Dysphagia and Cervical Spine Disorders in Patients With Neurologic Deficits Due to Brain Lesions
Brief Title: Dysphagia and Cervical Spine Disorders in Patients With Brain Lesions
Acronym: DysphagCerv
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Ioannina (Other)
Responsible Party: Principal Investigator, Avraam Ploumis, Assistant Professor of PMR, Orthopaedic Spine Surgeon, University of Ioannina
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 85/2010
Record Dates: First submitted 2011-07-28; First posted 2011-08-16 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Prevention; Rehabilitation
Keywords: spine injuries; brain lesions; dysphagia
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Videofluroscopic swallow study (VFSS) (Active Comparator): To investigate the swallowing ability of patients with neurologic problems
  Interventions: Procedure: Videofluroscopic swallow study (VFSS)
- cervical spine isometric excercises (Active Comparator): isometric exercises in patients with cervical spine scoliosis
  Interventions: Procedure: cervical spine isometric exercises
- Fiberoptic endoscopic esophageal study (FEES) (Active Comparator): To investigate the anatomic structures during swallowing of patients with neurologic problems
  Interventions: Procedure: Fiberoptic endoscopic esophageal study (FEES)

INTERVENTIONS:
Procedure: Videofluroscopic swallow study (VFSS) — Barium, radiation
  Arms: Videofluroscopic swallow study (VFSS)
Procedure: cervical spine isometric exercises — patients with cervical scoliosis will execute isometric exercises of the cervical spine
  Arms: cervical spine isometric excercises
Procedure: Fiberoptic endoscopic esophageal study (FEES) — food for swallowing
  Arms: Fiberoptic endoscopic esophageal study (FEES)

SUMMARY:
The research is about a prospective study conducted in patients suffering from dysphagia and cervical spine disorders and how they are interrelated. Three questionnaires have been given to patients with neurologic deficits, the first of these investigates the occurence of dysphagia in the three stages of swallowing, the second looks into the quality of life following a stroke or other neurologic damage and the third analyses how cervical spine disorders can affect every day life. After the bedside examination, VFSS or FEES, the patients are submitted to swallowing and cervical resistance exercises in fixed time periods after their hospitalisation. The results will be collected and evaluated using the statistical programme SPSS.

ELIGIBILITY:
Inclusion Criteria:

* brain lesions and cervical spine disorders

Exclusion Criteria:

* age
* peripheral damages

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2011-01; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
change in swallowing ability and quality of life by swal-quol questionnaire | at the time of admittance to the rehabilitation department (baseline), at six weeks, at one year
change of swallowing ability by Okuma's questionnaire | at the time of admittance to the rehabilitation department (baseline), at six weeks, at one year
change of cervical scoliosis measured by Cobb method in x-rays | at the time of admittance to the rehabilitation department (baseline), at six weeks, at one year

SECONDARY OUTCOMES:
change of cervical oswestry disability index | at the time of admittance to the rehabilitation department (baseline), at six weeks, at one year
  this questionnaire will be distributed only to patients with previous cervical spine problems

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Ioannina, Ioannina, Greece